CLINICAL TRIAL: NCT04539093
Title: Assessment of Endothelial Function in Patients With Advanced Heart Failure Requiring Mechanical Circulatory Support
Brief Title: Endothelial Function in Mechanical Circulatory Support
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Nicole Lohr, Associate Professor, Medical College of Wisconsin
Other Study IDs: PRO00038133
Record Dates: First submitted 2020-08-14; First posted 2020-09-04 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Endothelial Dysfunction; LVAD
Keywords: Observational; Pilot study

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Urine specimen - 1 sample per subject taken over a period of 1 day for urine pregnancy test. Up to a total of 60 (20 x 3 visits) samples for the duration of the project.
  Blood specimen - 1 sample per subject taken over a period of 1 day for measurement of blood nitric oxide levels. Up to a total of 60 (20 x 3 visits) samples for the duration of the project.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- End-stage heart failure patients requiring lvad support: Patients with end-stage heart failure with reduced ejection fraction, requiring mechanical circulatory support.
  Interventions: Other: Exposure of interest - Use of left ventricular assist device (LVAD)

INTERVENTIONS:
Other: Exposure of interest - Use of left ventricular assist device (LVAD) — Mechanical circulatory support devices such as left ventricular assist device is used as a treatment option for patients with end-stage heart failure.

SUMMARY:
The pathophysiology of HF is highly variable, with overlapping pathogenic mechanisms that complicates any attempt to create a simple and unified conceptual model. Left ventricular (LV) ejection fraction (EF), assessed as the fraction of the end-diastolic volume that is ejected upon contraction, has been the cornerstone metric for characterization of LV systolic function in patients with HF. LVEF demonstrates a strong inverse relationship with clinical outcomes in HF in patients with reduced EF (HFrEF). Current management options for the treatment of HFrEF include medical management, mechanical circulatory support, and cardiac transplantation. In the setting of refractory end stage HFrEF, the standard of care is heart transplantation. Since limited organ procurement is a significant constraint to the treatment of patients with advanced disease, durable mechanical circulatory support (MCS) with left ventricular assist devices (LVAD) were developed as a safe and efficacious treatment strategy for patients with advanced HF that is refractory to medical therapy.

The advances in LVAD engineering and design, tailored towards defined physiological goals, have resulted in the creation of much smaller continuous-flow (CF) pumps that possess technical superiority, pump durability, and ease of implantation compared to the older and larger pulsatile-flow pumps. The addition of speed modulation algorithms to the next generation centrifugal CF LVADs, has decreased the incidence of device related adverse events.

Our interest lies in the impact of continuous flow hemodynamics on endothelial function and the cardiac and end-organ responses to this novel therapy. Current knowledge of the impact of these specific advances in LVAD therapy is however limited by the relative youth of the field. Thus, the goal of this research project is to study human LVAD patients and to determine the impact of speed modulation algorithms in CF physiology on microvascular and endothelial function and its association with cardiac and peripheral organ function.

The investigators hypothesize that restoration of cardiac output using an LVAD with modern speed modulation algorithm improves vascular endothelial function. In addition, these changes would have a positive correlation with functional outcomes.

DETAILED DESCRIPTION:
The advances in LVAD engineering and design, tailored towards defined physiological goals, have resulted in the creation of much smaller CF pumps that possess technical superiority, pump durability, and ease of implantation compared to the older and larger PF pumps. The addition of artificial pulsatility to the next generation centrifugal CF LVADs, has decreased the incidence of device related adverse events. However, given the recent nature of these advances, the physiologic impact has yet to be fully elucidated. LVADs in general have demonstrated good outcomes and are rapidly gaining traction towards becoming standard therapy for refractory end stage HF. The investigators are in a position to study this new technology and the impact of the resultant altered physiologic state.

Our interest lies in the impact of continuous flow hemodynamics on endothelial function and the cardiac and end-organ responses to this novel therapy. Basal homeostatic properties of healthy endothelium are in part based on the effects of hemodynamic forces such as hydrostatic pressure, cyclic stretch, and fluid shear stress, which occur as a consequence of blood pressure and pulsatile blood flow in the vasculature. Under ambient conditions, these forces are generally atheroprotective and increase the expression of nitric oxide synthase (eNOS) to generate nitric oxide (NO), decrease reactive oxidative species (ROS) and oxidative stress, decrease expression of proinflammatory adhesion molecules, and maintain an antithrombotic surface. Increases in shear stress stimulate compensatory expansion of the vessels and thereby return shear forces to basal levels. Likewise, a decrease in shear stress can narrow the lumen of the vessel in an endothelium-dependent manner. In essence, the vessel remodels itself in response to long-term changes in flow, such that the luminal diameter is reshaped to maintain a constant predetermined level of shear stress. The capacity of the endothelium to sense shear stress is therefore an important determinant of luminal diameter and overall vessel structure. Failure to adapt to pathophysiological stimuli may lead to maladaptive responses that result in seemingly permanent alterations in endothelial phenotype and promote endothelial dysfunction. This phenomenon plays an integral role in several cardiovascular disease processes. Endothelial dysfunction (of both microvascular and conduit arteries) is a component of chronic heart failure and correlates with severity of disease. Improvement in cardiac function, whether via medical therapy or cardiac output augmentation, can improve endothelial function and benefit patients through better peripheral vascular reactivity. However, much of the improvement in endothelial function is thought to be related to the pulsatile laminar flow that occurs in majority of vascular beds. With the increasing use of CF pumps, it has become clear that the lack of pulsatility adversely affects the endothelium by decreasing vessel wall shear stress; reducing cyclic stretch that affects vascular cell proliferation; disrupting endothelium-dependent vasodilation; activating extrinsic pathway of thrombosis; and heightening vascular inflammation. The reintroduction of pulsatility through flow modulation control strategies could help mitigate these device specific issues and help promote endothelial recovery. Our knowledge of the impact of these specific advances in LVAD therapy is however limited by the relative youth of the field. Thus, the goal of this research project is to study human LVAD patients to determine the impact of artificial pulsatility in CF physiology on microvascular and endothelial function and its association with cardiac and peripheral organ function.

ELIGIBILITY:
Inclusion Criteria:

• Patients over the age of 18 years, deemed to be candidates for LVAD implantation. All ethnicities will be included in this study.

Exclusion Criteria:

* Age < 18 years or > 85 years.
* Presence of intra-cardiac shunt - safety concern for use of Echo contrast.
* Patient requiring temporary MCS - high acuity; may not be feasible to perform baseline assessment.
* Severe peripheral vascular disease - potential confounding bias during ultrasound assessment.
* Skeletal muscle disorder - not feasible to assess functional outcomes.
* Underlying/genetic vascular disease, i.e. vasculitis - potential for confounding bias during ultrasound assessment.
* Pregnant women - potential risk to fetus.
* Non-English Speaking.
* Active alcohol or illicit substance use.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End-stage heart failure patients at an academic medical center who are scheduled for LVAD implantation, will be screened for their candidacy in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of endothelial function | 9 months
  Measurement of blood nitric oxide levels will be used to evaluate vascular endothelial function. Flow-mediated dilation technique will then be used as a barometer of nitric oxide availability. The concentration of nitric oxide levels and degree of flow-mediated dilation would correlate with endothelial function.
Evaluation of microvascular function | 9 months
  Contrast enhanced ultrasound of the peripheral skeletal muscle of lower extremities will be used to evaluate microvascular function. Blood flow quantified using the ultrasound images would correlated with microvascular function.

SECONDARY OUTCOMES:
Functional outcomes - Quality of Life | 9 months
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item self-administered questionnaire that helps quantify the impact of heart failure on quality of life. This score will be used to determine correlations with endothelial function.
Functional outcomes - Mobility | 9 months
  The six-minute walk test (6MWT) is an index of physical function in patients with heart failure. The walking distance achieved by the 6MWT will be used to determine correlations with endothelial function.
Functional outcomes - Handgrip | 9 months
  Handgrip strength (HGS) measured by using a handheld dynamometer is a simple and effective means of assessing peripheral muscle strength. The degree of HGS will be used to determine correlations with endothelial function.
Functional outcomes - Lower extremity strength | 9 months
  The Five-repetition sit-to-stand test (FRSTST) is a widely used measure of lower extremity strength in clinical research and practice. The time taken to complete the test will be used to determine correlations with endothelial function.
Functional outcomes - Ventilation and gas exchange | 9 months
  The Cardiopulmonary Exercise Test (CPET) provides breath-by-breath gas exchange measures of 3 variables: O2 uptake (VO2), carbon dioxide output (VCO2), and ventilation (VE). These 3 measures will be used to determine correlations with endothelial function.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole L Lohr, MD PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided
Request not yet submitted to institution's Human Subject Protection Review Board.

REFERENCES:
- [Background] Mehra MR. The burden of haemocompatibility with left ventricular assist systems: a complex weave. Eur Heart J. 2019 Feb 21;40(8):673-677. doi: 10.1093/eurheartj/ehx036. No abstract available. PMID 28329374
- [Background] Kumar J, Elhassan A, Dimitrova G, Essandoh M. The Lavare Cycle: A Novel Pulsatile Feature of the HVAD Continuous-Flow Left Ventricular Assist Device. J Cardiothorac Vasc Anesth. 2019 Apr;33(4):1170-1171. doi: 10.1053/j.jvca.2018.11.029. Epub 2018 Nov 22. No abstract available. PMID 30630656
- [Background] Benjamin EJ, Muntner P, Alonso A, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Das SR, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Jordan LC, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, O'Flaherty M, Pandey A, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Spartano NL, Stokes A, Tirschwell DL, Tsao CW, Turakhia MP, VanWagner LB, Wilkins JT, Wong SS, Virani SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2019 Update: A Report From the American Heart Association. Circulation. 2019 Mar 5;139(10):e56-e528. doi: 10.1161/CIR.0000000000000659. No abstract available. PMID 30700139
- [Background] Essandoh M, Essandoh G, Stallkamp ED Jr, Perez WJ. Spectral Doppler Analysis of the HeartMate 3 Left Ventricular Assist Device Inflow: New Challenges Presented by the Artificial Pulse Technology. J Cardiothorac Vasc Anesth. 2018 Dec;32(6):e4-e5. doi: 10.1053/j.jvca.2018.07.005. Epub 2018 Jul 7. No abstract available. PMID 30108022
- [Background] Yost G, Bhat G. Relationship Between Handgrip Strength and Length of Stay for Left Ventricular Assist Device Implantation. Nutr Clin Pract. 2017 Feb;32(1):98-102. doi: 10.1177/0884533616665926. Epub 2016 Sep 25. PMID 27600398
- [Background] Steiner J, Wiafe S, Camuso J, Milley K, Wooster LT, Bailey CS, Thomas SS, D'Alessandro DA, Garcia JP, Lewis GD. Predicting Success: Left Ventricular Assist Device Explantation Evaluation Protocol Using Comprehensive Cardiopulmonary Exercise Testing. Circ Heart Fail. 2017 Jan;10(1):e003694. doi: 10.1161/CIRCHEARTFAILURE.116.003694. No abstract available. PMID 27998882
- [Background] Rogers JG, Pagani FD, Tatooles AJ, Bhat G, Slaughter MS, Birks EJ, Boyce SW, Najjar SS, Jeevanandam V, Anderson AS, Gregoric ID, Mallidi H, Leadley K, Aaronson KD, Frazier OH, Milano CA. Intrapericardial Left Ventricular Assist Device for Advanced Heart Failure. N Engl J Med. 2017 Feb 2;376(5):451-460. doi: 10.1056/NEJMoa1602954. PMID 28146651
- [Background] Mehra MR, Naka Y, Uriel N, Goldstein DJ, Cleveland JC Jr, Colombo PC, Walsh MN, Milano CA, Patel CB, Jorde UP, Pagani FD, Aaronson KD, Dean DA, McCants K, Itoh A, Ewald GA, Horstmanshof D, Long JW, Salerno C; MOMENTUM 3 Investigators. A Fully Magnetically Levitated Circulatory Pump for Advanced Heart Failure. N Engl J Med. 2017 Feb 2;376(5):440-450. doi: 10.1056/NEJMoa1610426. Epub 2016 Nov 16. PMID 27959709
- [Background] Dokainish H, Teo K, Zhu J, Roy A, AlHabib KF, ElSayed A, Palileo-Villaneuva L, Lopez-Jaramillo P, Karaye K, Yusoff K, Orlandini A, Sliwa K, Mondo C, Lanas F, Prabhakaran D, Badr A, Elmaghawry M, Damasceno A, Tibazarwa K, Belley-Cote E, Balasubramanian K, Islam S, Yacoub MH, Huffman MD, Harkness K, Grinvalds A, McKelvie R, Bangdiwala SI, Yusuf S; INTER-CHF Investigators. Global mortality variations in patients with heart failure: results from the International Congestive Heart Failure (INTER-CHF) prospective cohort study. Lancet Glob Health. 2017 Jul;5(7):e665-e672. doi: 10.1016/S2214-109X(17)30196-1. Epub 2017 May 3. PMID 28476564
- [Background] Bristow MR, Kao DP, Breathett KK, Altman NL, Gorcsan J 3rd, Gill EA, Lowes BD, Gilbert EM, Quaife RA, Mann DL. Structural and Functional Phenotyping of the Failing Heart: Is the Left Ventricular Ejection Fraction Obsolete? JACC Heart Fail. 2017 Nov;5(11):772-781. doi: 10.1016/j.jchf.2017.09.009. PMID 29096787
- [Background] Zimpfer D, Strueber M, Aigner P, Schmitto JD, Fiane AE, Larbalestier R, Tsui S, Jansz P, Simon A, Schueler S, Moscato F, Schima H. Evaluation of the HeartWare ventricular assist device Lavare cycle in a particle image velocimetry model and in clinical practice. Eur J Cardiothorac Surg. 2016 Nov;50(5):839-848. doi: 10.1093/ejcts/ezw232. Epub 2016 Sep 7. PMID 27605222
- [Background] Malhotra R, Bakken K, D'Elia E, Lewis GD. Cardiopulmonary Exercise Testing in Heart Failure. JACC Heart Fail. 2016 Aug;4(8):607-16. doi: 10.1016/j.jchf.2016.03.022. Epub 2016 Jun 8. PMID 27289406
- [Background] Lee M, Akashi H, Kato TS, Takayama H, Wu C, Xu K, Collado E, Weber MP, Kennel PJ, Brunjes DL, Ji R, Naka Y, George I, Mancini D, Farr M, Schulze PC. Vascular inflammation and abnormal aortic histomorphometry in patients after pulsatile- and continuous-flow left ventricular assist device placement. J Heart Lung Transplant. 2016 Sep;35(9):1085-91. doi: 10.1016/j.healun.2015.12.027. Epub 2016 Jan 6. PMID 26899764
- [Background] Schmitto JD, Hanke JS, Rojas SV, Avsar M, Haverich A. First implantation in man of a new magnetically levitated left ventricular assist device (HeartMate III). J Heart Lung Transplant. 2015 Jun;34(6):858-60. doi: 10.1016/j.healun.2015.03.001. Epub 2015 Mar 7. No abstract available. PMID 25920932
- [Background] Moazami N, Dembitsky WP, Adamson R, Steffen RJ, Soltesz EG, Starling RC, Fukamachi K. Does pulsatility matter in the era of continuous-flow blood pumps? J Heart Lung Transplant. 2015 Aug;34(8):999-1004. doi: 10.1016/j.healun.2014.09.012. Epub 2014 Sep 28. PMID 25447568
- [Background] Matsuzawa Y, Kwon TG, Lennon RJ, Lerman LO, Lerman A. Prognostic Value of Flow-Mediated Vasodilation in Brachial Artery and Fingertip Artery for Cardiovascular Events: A Systematic Review and Meta-Analysis. J Am Heart Assoc. 2015 Nov 13;4(11):e002270. doi: 10.1161/JAHA.115.002270. PMID 26567372
- [Background] Ising MS, Sobieski MA, Slaughter MS, Koenig SC, Giridharan GA. Feasibility of Pump Speed Modulation for Restoring Vascular Pulsatility with Rotary Blood Pumps. ASAIO J. 2015 Sep-Oct;61(5):526-32. doi: 10.1097/MAT.0000000000000262. PMID 26102173
- [Background] Watanabe A, Amiya E, Hatano M, Watanabe M, Ozeki A, Nitta D, Maki H, Hosoya Y, Tsuji M, Bujo C, Saito A, Endo M, Kagami Y, Nemoto M, Nawata K, Kinoshita O, Kimura M, Ono M, Komuro I. Significant impact of left ventricular assist device models on the value of flow-mediated dilation: effects of LVAD on endothelial function. Heart Vessels. 2020 Feb;35(2):207-213. doi: 10.1007/s00380-019-01474-2. Epub 2019 Jul 20. PMID 31327031
- [Background] Symons JD, Deeter L, Deeter N, Bonn T, Cho JM, Ferrin P, McCreath L, Diakos NA, Taleb I, Alharethi R, McKellar S, Wever-Pinzon O, Navankasattusas S, Selzman CH, Fang JC, Drakos SG. Effect of Continuous-Flow Left Ventricular Assist Device Support on Coronary Artery Endothelial Function in Ischemic and Nonischemic Cardiomyopathy. Circ Heart Fail. 2019 Aug;12(8):e006085. doi: 10.1161/CIRCHEARTFAILURE.119.006085. Epub 2019 Aug 19. PMID 31422672
- [Background] Hydren JR, Kithas AC, Park SH, Wever-Pinzon O, Selzman CH, Perry W, Vargas CAS, Stehlik J, Drakos SG, Richardson RS. Targeting Peripheral Vascular Pulsatility in Heart Failure Patients with Continuous-Flow Left Ventricular Assist Devices: The Impact of Pump Speed. ASAIO J. 2020 Mar;66(3):291-299. doi: 10.1097/MAT.0000000000001001. PMID 30973399
- [Background] Witman MA, Garten RS, Gifford JR, Groot HJ, Trinity JD, Stehlik J, Nativi JN, Selzman CH, Drakos SG, Richardson RS. Further Peripheral Vascular Dysfunction in Heart Failure Patients With a Continuous-Flow Left Ventricular Assist Device: The Role of Pulsatility. JACC Heart Fail. 2015 Sep;3(9):703-11. doi: 10.1016/j.jchf.2015.04.012. Epub 2015 Aug 12. PMID 26277768
- [Background] Amir O, Radovancevic B, Delgado RM 3rd, Kar B, Radovancevic R, Henderson M, Cohn WE, Smart FW. Peripheral vascular reactivity in patients with pulsatile vs axial flow left ventricular assist device support. J Heart Lung Transplant. 2006 Apr;25(4):391-4. doi: 10.1016/j.healun.2005.11.439. Epub 2006 Feb 3. PMID 16563966
- [Background] Corretti MC, Anderson TJ, Benjamin EJ, Celermajer D, Charbonneau F, Creager MA, Deanfield J, Drexler H, Gerhard-Herman M, Herrington D, Vallance P, Vita J, Vogel R; International Brachial Artery Reactivity Task Force. Guidelines for the ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery: a report of the International Brachial Artery Reactivity Task Force. J Am Coll Cardiol. 2002 Jan 16;39(2):257-65. doi: 10.1016/s0735-1097(01)01746-6. PMID 11788217
- [Background] Leeson P, Thorne S, Donald A, Mullen M, Clarkson P, Deanfield J. Non-invasive measurement of endothelial function: effect on brachial artery dilatation of graded endothelial dependent and independent stimuli. Heart. 1997 Jul;78(1):22-7. doi: 10.1136/hrt.78.1.22. PMID 9290397
- [Background] Khan T, Levin HR, Oz MC, Katz SD. Delayed reversal of impaired metabolic vasodilation in patients with end-stage heart failure during long-term circulatory support with a left ventricular assist device. J Heart Lung Transplant. 1997 Apr;16(4):449-53. PMID 9154956